CLINICAL TRIAL: NCT02609932
Title: Effect of Interferon-gamma 1-b on Innate Immune Cells
Brief Title: Effect of IFN-γ on Innate Immune Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-1643; UL1TR001082 (NIH)
Record Dates: First submitted 2015-11-11; First posted 2015-11-20 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Chronic Granulomatous Disease
Keywords: Interferon-gamma; innate immunity
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — Interferon-gamma; interferon gamma-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SD or SS (Other): In this study, IFN- γ-1b will be subcutaneously administered a total of 30 subjects in one of two cohorts; Single Dose (SD) or Steady State (SS) dosing. Dosing of IFN- γ-1b will be based upon the time subject became eligible and started study. In this non-randomized, open-label study, subjects will be enrolled on the SD cohort first, and once that cohort has been filled, enrollment to the SS cohort will begin. Although not required, subjects in the SD cohort may also volunteer to participate in the SS cohort if they still meet eligibility criteria. Separate consents will be used for the SD and SS cohorts. In the event not all the SD subjects choose to continue onto the SS cohort, we will plan to recruit new participants from our local campus community.
  Interventions: Drug: Administration of drug (Interferon-gamma 1-b) subcutaneously

INTERVENTIONS:
Drug: Administration of drug (Interferon-gamma 1-b) subcutaneously — SD = group who has received a single dose of IFN-gamma (10, 25, 50, and 100 mcg/m2) given once with subsequent analysis of effects (serum IL-10, Neuropterin, and IFN levels as well as neutrophil Nox2 activity and gene expression by Affimetrics Chip analysis). One month is allowed between doses. SS = administration of four doses (50 mcg/m2) of IFN-gamma given on Monday, Wednesday Friday schedule with neutrophil or monocyte function studies performed before the first and after the fourth dose to determine steady state effects.
  Other Names: Actimmune

SUMMARY:
The investigators hypothesize that neutrophils and monocytes developed under the influence of Interferon- gamma-1b (IFN-γ-1b, Actimmune*) in vivo will display enhanced function across a broad range of activities related in large part to the transcriptional activation effects of this cytokine. The investigators will evaluate the effects of IFN-γ in healthy human subjects in vivo on gene expression, biologic activity markers, and functional activity of myeloid cells in single dose studies and in steady state studies.

DETAILED DESCRIPTION:
Named for their potent ability to interfere and protect against viral infections, interferons (IFNs) have many regulatory effects on the immune system.1 Of the members of the two classes of these compounds, IFN-γ has the most diverse and powerful immune effects. Studies have mostly evaluated IFN-γ interactions with cells of adaptive immunity, including macrophages and lymphocytes. Effects on innate immunity, particularly polymorphonuclear leukocytes or neutrophils and monocytes are less well studied. However, investigations have suggested that IFN-γ may be involved in signal transduction, gene expression, the respiratory burst and neutrophil NADPH oxidase (Nox2) activity, phagocytosis, motility, microbicidal activity, and apoptosis. Not all of these functions are enhanced by IFN-γ; but the clinical use of this cytokine has been driven, in part by these results. For example, the primary motivation for initiating investigation of its beneficial clinical effects in Chronic Granulomatous Disease (CGD) was its effects on Nox2 activity.2 Most data in this area was based on studies using differentiated neutrophils from peripheral blood.1 However, the phenotype of neutrophils developed under the influence of this cytokine, not just changes expressed by exposure of differentiated cells to IFN-γ, is critical to understanding the physiologic effects of IFN-γ and the broad applications for its use in treatment of a range of human diseases. To expand their understanding of the role of IFN-γ in the development and functional integrity of the neutrophil, the investigators have completed a series of studies with PLB-985 cells in an in vitro culture system of myeloid cells. In this proposal, the investigators will evaluate innate immune activation and phagocyte function in healthy adult volunteers who are receiving IFN-γ.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults over the age of 18 years up to 60 years.
2. At time of screening subject is well and healthy;
3. Acute infections resolved;
4. Subject off treatment medications;
5. No diagnosis of chronic conditions or active health care issues for which the subject is actively followed by a health care provider or is on chronic medications.
6. Non-prescription medications for mild inter-current illnesses will be allowed at the discretion of the principal investigator.

Exclusion Criteria:

1. Pregnancy.
2. History of current infection;
3. Two weeks from most recent intercurrent infection;
4. History of recurrent infections or immunodeficiency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2018-08 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in Neutrophil Nox2 activity. | Determine the change in Nox2 activity at baseline compared to results for 8,24,48,72,96 hours after each IFN dose for the SD cohort.
  Nox2 activity will be measured by DHR oxidation or Sod inhibitable cytochrome c reduction.
Change in Plasma IL-10 and Neuropterin concentration. | Determine the change in IL-10 and neuropterin concentration at baseline compared to 4, 8, 12, 24, 36, 48, 72, and 96 hours after each IFN dose, SD cohort.
  IL-10nd Neuropterin will be measured by ELISA.
Change in Neutrophil Gene Expression Analysis. | Determine the change in gene expression at baseline compared to 4, 8, 12, 24, 36, 48, 72, and 96 hours after each IFN dose, SD cohort.
  RNA will be extracted and gene expression will be determined by Affimetrix Gene Chip assay.
Change in IFN concentration and detection of anti-IFN antibody | Determine the change in IFN level at baseline compared to 4, 8, 12, and 24 hours after administration of each dose of IFN-gamma in the SD cohort. Determine the change in IFN antibody at baseline compared to day 7-10 and day 30 after IFN
  IFN levels and anti-drug antibody will be completed by standard assays.

SECONDARY OUTCOMES:
Change in Neutrophil Function studies. | Determine the change in neutrophil function at baseline compared to results on Day 8 after the 4th dose of IFN.
  Neutrophil chemotaxis, bactericidal activity,ingestion, degranulation, f-Actin expression, CD11b/18 expression, Nox2 activity to a variety of agonists.
Change in Anti-IFN antibody. | Determine the change in IFN antibody at baseline compared to results for 7-10 da. and 30 da. after IFN.
  Anti-drug antibody to be determined by standard assay.
Change in Monocyte function studies. | Determine the change in monocyte function at baseline compared to results on Day 8 after the 4th dose of IFN.
  Monocyte chemotaxis, bactericidal activity,ingestion, Expression of monocyte specific surface determinants, CD11b/18 expression, Nox2 activity to a variety of agonists, cell content of specific proteins, and antibody dependent cellular cytotoxicity.
Change in Neutrophil and Monocyte Gene Expression Analysis. | Determine the change in monocyte function at baseline compared to results on Day 8 after the 4th dose of IFN.
  RNA will be extracted and gene expression will be determined by Affimetrix Gene Chip assay.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R. Ambruso, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellison MA, Thurman G, Gearheart CM, Seewald RH, Porter CC, Ambruso DR. INF-gamma Enhances Nox2 Activity by Upregulating phox Proteins When Applied to Differentiating PLB-985 Cells but Does Not Induce Nox2 Activity by Itself. PLoS One. 2015 Aug 28;10(8):e0136766. doi: 10.1371/journal.pone.0136766. eCollection 2015. PMID 26317224
- [Derived] Ambruso DR, Briones NJ, Baroffio AF, Murphy JR, Tran AD, Gowan K, Sanford B, Ellison M, Jones KL. In vivo interferon-gamma induced changes in gene expression dramatically alter neutrophil phenotype. PLoS One. 2022 Feb 3;17(2):e0263370. doi: 10.1371/journal.pone.0263370. eCollection 2022. PMID 35113934